CLINICAL TRIAL: NCT06002815
Title: Comparison of Nasogastric Tube Insertion Success in Difficult and Easy Airway Patients
Status: Completed | Type: Observational
Sponsor: Taksim Egitim ve Arastirma Hastanesi (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023.07.IRB.78
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to investigate potential variations in the success rate and occurrence of complications during nasogastric tube insertion between Difficult and Easy Airway Patients.

DETAILED DESCRIPTION:
Patients who are scheduled for surgery for any reason and who will receive general anesthesia requiring perioperative nasogastric tube insertion will be included in the study. Two groups will be formed, the easy airway group and the difficult airway group. The main aim is to investigate whether there is a difference between the groups in terms of the success of insertion of the nasogastric tube (first attempt, second attempt etc.) and the duration of insertion. Investigating the differences between the groups in terms of complications such as bleeding, twisting in the mouth, kinking, and going to the trachea is determined as a secondary aim. At the end of the study, determining the correlation between the failure of nasogastric tube insertion and difficult airway parameters is planned as another secondary goal.

ELIGIBILITY:
Inclusion Criteria: Patients who are scheduled for surgery for any reason and who will receive general anesthesia requiring perioperative nasogastric tube insertion will be included in the study.

-

Exclusion Criteria:

* Patients under 18 year-old
* Patients who do not require nasogastric tube insertion
* Patients with anatomical changes in the head and neck region
* Patients without an informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for surgery for any reason and who will receive general anesthesia requiring perioperative nasogastric tube insertion will be included in the study.
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Comparison of Nasogastric Tube Insertion in Difficult and Easy Airway Patients | 10 minutes
  The main aim was to investigate whether there is a difference between the groups in terms of the success of insertion of the nasogastric tube (first attempt, second attempt etc.) and the duration of insertion

SECONDARY OUTCOMES:
Complications in Difficult and Easy Airway Patients | 5 minutes
  Investigating the differences between the groups in terms of complications such as bleeding, twisting in the mouth, kinking, and going to the trachea is determined as a secondary aim
Airway parameters and failure of nasogastric tube insertion | 10 minutes
  Determining the correlation between the failure of nasogastric tube insertion and difficult airway parameters is planned as another secondary goal.

CONTACTS AND LOCATIONS:
Overall Officials: Celal Kaya, MD, Principal Investigator — Taksim Training and Research Hospital
Locations (1):
- Taksim Training and Research Hospital, Istanbul, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.